CLINICAL TRIAL: NCT00937885
Title: Consequences From Use of Reminiscence: a Randomised Intervention Study in Ten Danish Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Nørrebro Erindringscenter - the Danish Centre for Reminiscence (Unknown); VIA University College (Other)
Responsible Party: Charlotte Horsted, CAST - Centre for Applied Health Services Research & Technology Assessment
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-41-4870
Record Dates: First submitted 2009-07-07; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Consequences for Nursing Home Residents and Staff of Integrating Reminiscence Into Daily Nursing Care.
Keywords: Reminiscence; Nursing home staff; Nursing home residents; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Implementation of reminiscence (Experimental): Individual and group reminiscence sessions held with residents, supplemented by reminiscence boxes, posters and exhibitions.
  Interventions: Behavioral: Implementation of reminiscence
- Usual nursing care (No Intervention)

INTERVENTIONS:
Behavioral: Implementation of reminiscence
  Arms: Implementation of reminiscence

SUMMARY:
Reminiscence is the systematic use of memories and recollections to strengthen self-identity and self-worth. The study aim was to investigate the consequences for nursing home residents and staff of integrating reminiscence into daily nursing care. Ten nursing homes were randomised into either an Intervention Group, who implemented reminiscence, or a Control Group, who continued with usual care. Data were collected at baseline and again 6 and 12 months after the intervention start. Results suggested that use of reminiscence can improve residents' quality of life and possibly delay progression in dementia symptoms. Nursing staff can experience greater satisfaction with personal and professional roles and develop a more positive view of the residents.

ELIGIBILITY:
Inclusion Criteria:

* nursing homes in the Mid-Jutland Region with at least one 35 residents who were willing to particpate in study
* signed informed consent from residents/relatives

Exclusion Criteria:

* nursing homes that already used reminiscence on a systematic basis
* nursing homes with recent organisational changes/extensive staff training
* residents in protected-environment units, were bed-ridden/terminally ill or on short-term placement.

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Nurses' attitudes towards professional role and contact with residents | 1 year

SECONDARY OUTCOMES:
Residents' quality of life (proxy assessment) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CAST - Centre for Applied Health Services Research & Technology Assessment, University of Southern Denmark, Odense, Denmark